Current Version: AMENDMENT #3: 2018-OCT-31

CONSENT FORM DATE: 2015-JUL-24

CCTG TRIAL: SC.24

AMEND #1: 2017-FEB-02

#### SAMPLE Informed Consent Form

A RANDOMIZED PHASE II/III STUDY COMPARING STEREOTACTIC BODY RADIOTHERAPY (SBRT) VERSUS CONVENTIONAL PALLIATIVE RADIOTHERAPY (CRT) FOR PATIENTS WITH SPINAL METASTASES

| TON FATILITIS WITH SEINAL WILLIASTASES |
|---|
| Trial Code: SC.24 |
| Study Doctor: Dr |
| Sponsor: Canadian Cancer Trials Group |
| Le formulaire de consentement est disponible en français sur demande. |
| Note: If an REB approved French consent is not used at your institution you should remove the above statement. |
| Emergency Contact Number (24 hours / 7 days a week): |
| Non-Emergency contact numbers are noted at the end of this document under the section neading "Contacts". |

# **INTRODUCTION**

You are being invited to participate in a clinical trial (a type of study that involves research). Clinical trials only include participants who choose to take part. You are invited to participate in this trial because you have cancer that has spread to your spine, called "spinal metastases", and it is causing you to have pain. This consent form provides you with information to help you make an informed choice. Please read this document carefully and take your time in making your decision. You may find it helpful to discuss it with your friends and family.

Taking part in this study is voluntary. You may choose not to take part or if you choose to participate may leave the study at any time without giving a reason. Deciding not to take part or deciding to leave the study later will not result in any penalty or any loss of benefits to which you are entitled.

### **BACKGROUND**

The standard or usual treatment to help reduce the pain in your spine is 'conventional radiation therapy' or CRT which provides a 'standard' dose of radiotherapy. This treatment is often effective in reducing pain, but may not get rid of the pain completely. Also, pain may return, even after the CRT has initially been effective.

Stereotactic Body Radiation Therapy or SBRT is a new form of radiation therapy which is able to deliver high doses of radiation to the specific painful area of your spine most affected by cancer. Special protective procedures and steps are taken to keep the radiation beams away from the healthy parts of your body that surround the cancer. The aim of delivering high doses of radiation is to help control the cancer and, in doing so, allow for better pain relief. But it is not clear if SBRT can offer better pain relief results than the standard treatment CRT.

CCTG TRIAL: SC.24

AMEND #1: 2017-FEB-02; AMEND #2: 2018-APR-03; AMEND #3: 2018-OCT-31 The research ethics board, which oversees the ethical conduct of research involving humans, has reviewed and accepted this study.

### **PURPOSE**

The purpose of this study is to find out if SBRT is better than CRT at controlling pain in the spine 3 months after receiving treatment. The first part of the randomized trial (phase II) looked at whether it was possible (feasible) to provide these treatments in cancer centres across Canada, by aiming to recruit 54 participants within 18 months. This part of the study was successfully completed in early 2017. Participants of this feasibility stage of the study will not need to have any extra procedures than originally planned.

The next stage, called a randomized **phase III** trial, is now underway. It involves recruiting another 174 participants to receive either CRT or SBRT, using exactly the same study procedure as in the feasibility study. We will continue to obtain information about whether SBRT is better than CRT at controlling pain.

This research is being done because while there is some evidence suggesting that SBRT may improve treatment for patients with spine metastases, more research is needed to determine if it is better than CRT. This increase to a total of 228 study participants will help investigators to answer the study question.

### ALTERNATIVE TREATMENTS

You do not have to take part in this study in order to receive treatment/care. Other options (in addition to the standard or usual treatment described above) may include, but are not limited to:

- no therapy at this time
- the standard radiation therapy, CRT
- you may be able to get study treatment, SBRT, at this centre or other centres (if they have the ability to deliver the treatment) even if you do not take part in the study.
- palliative care or Best Supportive Care (BSC). This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Best Supportive Care tries to keep you as active and comfortable as possible.
- other experimental studies may be available if you do not take part in this study

Please talk to your study doctor or usual cancer doctor about the known benefits and risks of these other options before you decide to take part in this study. Your usual cancer doctor can also discuss with you what will happen if you decide not to undertake any treatment at this time.

# **EXPECTED NUMBER OF PARTICIPANTS**

Up to 228 people will take part in this study in Canada and Australia. The study should take 4 years to complete and the results should be known approximately 1 year later.

Your study doctor will be informed of the results of this study once they are known.

CCTG TRIAL: SC.24

### ASSIGNMENT TO A GROUP

If you decide to participate then you will be "randomized" into one of the groups described below. Randomization means that you are put into a group by chance (like flipping a coin). There is no way to predict which group you will be assigned to. You will have an equal chance of being placed in either group. Neither you nor your study doctor can choose what group you will be in.

You will be told which treatment you are to get.

### **EXPERIMENTAL TREATMENT:**

# Group 1 (STANDARD TREATMENT): Conventional Radiation Therapy (CRT)

If you are randomized to Group 1 you will receive standard doses of radiation given as one treatment per day for five days. This treatment is referred to as 'conventional radiation therapy' or CRT. To prepare for your radiation treatment, you will first have a planning procedure. This involves having a CT scan (a special X-ray) to map the area of your spine that is to receive radiation. The images from the CT scan will be used to determine where the treatment beams from the radiation machine should be directed.

# **Group 2** (NEW TREATMENT): Stereotactic Body Radiotherapy (SBRT)

If you are randomized to Group 2 you will receive higher doses of radiation given as one treatment per day for two days. This new treatment is referred to as stereotactic body radiation therapy (SBRT). To prepare for your radiation treatment, you will first have two planning procedures. These involve having a CT scan (a special X-ray) and an MRI scan to map the area of your spine that is to receive radiation. The images from the CT and MRI scans will be used to determine where the treatment beams from the radiation machine should be directed. A main difference between SBRT and CRT is that with SBRT, you will be immobilized (your movement will be limited) in a special body immobilization device, or a special mask if your tumor is in the neck or upper back, for about 1 hour for each treatment. These devices will also be used when you have your CT scan that will be used to plan your radiation treatment and during your radiation treatment. The reason for using these devices is to make you as secure as possible and ensure you do not move during treatment.

# **STUDY PROCEDURES**

#### Non-Experimental Procedures

The following tests will be done as part of this study. Some of these tests may be done as part of your standard care, in which case the results may be used. Some of these tests may be done more frequently than if you were not taking part in this study and some may be done solely for the purpose of the study. If the results show that you are not able to continue participating, your study doctor will let you know.

- physical examination
- pregnancy test

AMEND #2: 2018-APR-03

magnetic resonance imaging (MRI) of the spine – a scan that uses a strong magnet to
produce pictures of areas inside the body such as organs and other tissue, and inside of
bones. In this case, the MRI of the spine will be done first to make sure that you are eligible
for this study. MRIs of your spine will also be done after you are enrolled on this study, to
allow the doctors to plan your radiotherapy treatment, and also to see if the cancer in your
spine is getting worse or not.

#### Questionnaires

This study has a Quality of Life and a Health Economics Questionnaire. The purpose of the questionnaires is to understand how your treatment and illness affects your quality of life, to understand how important different aspects of your health are to you and the costs associated with the treatments and your illness.

You will be provided with the questionnaire before enrolling on this study, on the first day that your radiotherapy is to be given to you, but *prior* to receiving this treatment, and then at 4 weeks and 3 and 6 months after the end of the radiotherapy study treatment. Each questionnaire will take about 10 minutes to complete.

You will complete the questionnaires electronically using a system called ePRO or using a paper based form if ePRO is not available at the centre where you are treated. Study personnel will explain how to complete the questionnaires. Tablet computers running the ePRO system will be kept at the clinic. If you have any questions about the completing of the questionnaire, please contact the study personnel listed below, during office hours.

The information you provide is for research purposes only and will remain strictly confidential. Some of the questions are personal; you can choose not to answer these if you wish.

Even though you may have provided information on a questionnaire, these responses may or may not be reviewed by your health care team or study team - if you wish them to know this information please bring it to their attention.

### **Participant Diary**

For this study, you will also need to keep a diary to tell the researchers how much pain you are having and how much medication you are taking to treat your pain. You will fill out the Patient Diary before enrolling on this study, on the first day that your radiotherapy is to be given to you, but *prior* to receiving this treatment, and then at 4 weeks and 3 and 6 months after the end of the radiotherapy study treatment. You will be asked to return the diary to the clinic/hospital.

You must be able to fill out the diary to participate on this study.

CCTG TRIAL: SC.24

AMEND #2: 2018-APR-03

# Central Radiology Review

Copies of your MRI images, at the time of study entry, as well as at 3 and 6 months after the end of radiotherapy, will be collected electronically as part of this study. This is required for quality assurance and data management. The electronic copies will be uploaded to a webbased, password-protected system, where they will be accessed by a designated study reviewer, based in one of the Canadian centres participating in this study. The images will be stored indefinitely.

To protect your identity, the information that will be on your MRI scans will be limited to study identifiers, such as your study code and initials.

# Central Radiotherapy Review

Copies of records providing information about the radiotherapy (SBRT or CRT) you will receive on this study, will be collected electronically. This is required for quality assurance and data management. The electronic copies will be uploaded to a web-based, password-protected system, where they will be accessed by a designated study reviewer, based in one of the Canadian centres participating in this study. These records will be stored indefinitely.

To protect your identity, the information that will be on your documentation will be limited to study identifiers, such as your study code and initials.

# Optional Sample Collection and Banking

The researchers doing this study are interested in doing additional research now or in the future on blood samples collected from you. You will be given an additional optional study consent form to read and sign if you wish to give permission for the blood samples to be banked (stored) for future research purposes. You may decide not to participate in the "optional" study and still participate in this main study.

# **RESPONSIBILITIES**

If you choose to participate in this study, you will be expected to:

- Tell your study doctor about your current medical conditions;
- Tell your study doctor if you are thinking about participating on another research study.
- Return any diaries or questionnaires that were completed to the clinic/hospital.
- Tell your study doctor if you become pregnant or father a child while participating on this study.

#### LENGTH OF PARTICIPATION

Your treatment will last for 5 days if you are randomized to Group 1 (CRT). If you are randomized to Group 2 (SBRT) your treatment will last for 2 days.

AMEND #1: 2017-FEB-02; AMEND #2: 2018-APR-03

You will be asked to come back to the clinic/hospital 4 weeks after the last dose of study treatment. You will then be asked to come back 3 and 6 months after the last dose of study treatment.

You may be seen more often if your study doctor determines that this is necessary, or if your cancer gets worse.

**Note**: indicate the overall length of time required beyond that of the standard or usual care - specifying the difference in the number of visits and the length of time for each visit plus the time needed to complete questionnaires or diaries.

No matter which group you are randomized to, and even if you stop treatment early, we would like to keep track of your health for 6 months after the last dose of study radiotherapy to look at the long-term effects of your participation on this study. We would do this by contacting you in person and/or asking you to come to the clinic 4 weeks, 3 months and 6 months after you receive the last dose of study radiotherapy.

# **EARLY END TO PARTICIPATION**

Your participation in the trial may be stopped early, for reasons such as:

- You are unable to tolerate the study treatment.
- New information shows that the study treatment is no longer in your best interest.
- Your study doctor no longer feels this is the best treatment for you.
- Canadian Cancer Trials Group (CCTG) decides to stop the study.
- If you become pregnant.

If your participation in the study is stopped your study doctor will provide information about how to stop safely.

#### RISKS OF PARTICIPATION

Participating in this study will put you at risk for the side effects listed below. You should discuss these with your study doctor. As with any treatment additional unexpected and sometimes serious side effects are a possibility.

Your study doctor will watch you closely to see if you have side effects. When possible, other drugs will be given to you to make side effects less serious and more tolerable. Many side effects go away shortly after your treatment is stopped but in some cases side effects can be serious, long-lasting, permanent, or may even cause death.

If you experience serious side effects that require treatment between regular clinic/hospital visits, it is important that you make every effort to return to the clinic/hospital where study radiotherapy was given. Because SBRT is a new radiotherapy technique and is only used in clinics/hospitals involved in research studies, any serious side effects may be best treated by these clinics/hospitals. If you need immediate treatment and are unable to return to the clinic/hospital where study radiotherapy was given, you should go to the nearest medical clinic/hospital and tell them that your study doctor should be contacted as soon as possible.

CCTG TRIAL: SC.24

Risks and side effects related to the <u>STEREOTACTIC BODY RADIOTHERAPY</u> we are studying include

Very likely (21% or more, or more than 20 people in 100):

- fatigue
- soreness
- pain flare. This means that the pain you have already that is caused by your disease has gotten slightly worse. This could also refer to development of new pain that you begin to experience after you completed your treatment.
- · skin redness in the area being treated
- damage to organs in the area receiving radiotherapy
- dry throat

# Less likely (5– 20% or between 5 and 20 people in 100):

- changes in how temperature is experienced
- weakness and clumsiness on one or both sides of the body
- episodes of pain or electric shock sensations down your back or legs

# Rarely (1 - 4% or less than 5 in 100 people):

 Vertebral compression fracture. This means that one of the small bones in your backbone has broken and as a result your backbone has shortened. This risk may be greater with SBRT than with CRT.

### Very Rarely (less than 1%):

 Damage to the spinal cord from radiation (called radiation myelopathy). This can be very serious as spinal cord injury can leave you paralyzed (loss of function) or can cause you to lose your bladder and bowel functions. This risk may be greater with SBRT than with CRT.

The risks and side-effects of the standard or usual treatment will be explained to you as part of your standard care and are therefore not listed.

Long term effects of the radiation used in this study include an increased risk of developing other cancers.

### REPRODUCTIVE RISKS

Radiotherapy may harm an unborn baby (fetus). You must not become pregnant or father a baby while receiving treatment and for 6 months after the last dose. Your study doctor will discuss methods with you to ensure that you do not become pregnant or father a baby during the study.

If you become pregnant or father a child during this study or for 6 months after the end of study treatment, then you should immediately notify your study doctor. Your study doctor will let the sponsor know about the pregnancy.

AMEND #1: 2017-FEB-02; AMEND #2: 2018-APR-03

If you become pregnant, the researchers or sponsors for this study will access information on the outcome of the pregnancy. This information will be gathered from your medical/study record. This may also involve contacting you for the next one year to ask about the health of your child. We may also ask to contact the child's father to get information related to the pregnancy. If you become pregnant and do not want the researchers/sponsors to collect this information, you must let your study doctor know.

If you father a child, the researchers or sponsor for this study will ask to contact the child's mother to collect information on the outcome of the pregnancy (the child's health, etc.). Your partner will be given a separate consent document to sign to give permission for the collection of this information, if a pregnancy should happen. Your partner may choose not to give consent for the collection of this information or may withdraw their consent at any time without giving a reason. This will not impact your participation on the study and will not result in any penalty or any loss of benefits to which you are entitled.

Radiotherapy used in this study may make you unable to have children in the future. Your study doctor will discuss this with you.

#### DATA SAFETY MONITORING BOARD

A Data Safety Monitoring board, an independent group of experts, will be reviewing the data from this research throughout the study.

#### **BENEFITS**

If you agree to take part in this study, SBRT may or may not be of direct benefit to you. We hope the information learned from this study will help other patients in the future.

# CONFIDENTIALITY

**Note:** If there will be a disclosure of personal identifiers i.e. disclosed on research-related information/documents, including samples and scans or as part of the unique identifier, - these disclosures must be justified in the REB application and approved. Please ensure that you are aware of all institutional and REB policies with respect to the disclosure of personal identifiers; specifically date of birth and initials. If the REB or institution mandates the disclosure only of partial date of birth (year/month), and/or of scrambled/coded initials, this will be accepted.

Records identifying you at this centre will be kept confidential and, to the extent permitted by the applicable laws, will not be disclosed or made publicly available, except as described in this consent document.

Authorized representatives of the following organizations may **look** at your original (identifiable) medical/clinical study records at the site where these records are held, for quality assurance (to check that the information collected for the study is correct and follows proper laws and quidelines).

- Canadian Cancer Trials Group (CCTG), the research group coordinating this study
- The research ethics board which oversees the ethical conduct of this study in your clinic/hospital.

Authorized representatives of the above organizations and the parties listed below may <u>receive</u> information related to the study from your medical/clinical study records for quality assurance and data analysis. Your name or other information that may identify you will not be used. The records received by these organizations may contain your participant code and initials.

- The central review centre (Odette Cancer Centre Sunnybrook Health Sciences Centre) located in Toronto, which will review the MRI spine images, so as to determine how the cancer in your spine responded to your study treatment
- The central review centre (Odette Cancer Centre Sunnybrook Health Sciences Centre), located in Toronto, which will review the radiotherapy documentation, to make sure that you received study treatment appropriately

All of the organizations listed in the above confidentiality sections are required to have strict policies and procedures to keep the information they see or receive about you confidential, except where disclosure may be required by law. The study doctor will ensure that any personal health information collected for this study is kept in a secure and confidential location as required by law. There are federal and provincial laws that these organizations must comply with to protect your privacy.

If the results of this study are published, your identity will remain confidential. It is expected that the information collected during this study will be used in analyses and will be published/presented to the scientific community at meetings and in journals.

Even though the likelihood that someone may identify you from the study data is very small, it can never be completely eliminated.

A copy of this signed and dated consent form may be included in your health record/hospital chart.

Your family doctor/health care provider will be informed that you are taking part in a study so that you can be provided with appropriate medical care. If you do not want you family doctor/health care provider to be informed, please discuss with your study doctor.

## REGISTRATION OF CLINICAL TRIALS

A description of this clinical trial will be available on <a href="www.clinicaltrials.gov">www.clinicaltrials.gov</a>. This website will not include information that can identify you. You can search this website at any time.

#### COSTS

The study treatment (radiotherapy) will be given to you free of charge.

The costs of your medical treatment will be paid for by your provincial medical plan to the extent that such coverage is available. There may be extra costs that are not covered by your medical plan that you will have to pay yourself, some examples may be physiotherapy or certain pain medications.

AMEND #1: 2017-FEB-02; AMEND #2: 2018-APR-03

Taking part in this study may result in added costs to you (i.e. transportation, parking, meals, or unpaid leave from work). You may have to pay for medication prescribed to treat or prevent side effects, and you may have to visit the hospital more often than if you were not participating in this study.

### COMPENSATION

You will not be paid for taking part in this study.

In the case of research-related side effects or injury, medical care will be provided by your doctor or you will be referred for appropriate medical care.

#### **RIGHTS**

You will be told, in a timely manner, about new information that may be relevant to your willingness to stay in this study.

If you decide to stop participating in the study or if your participation has been stopped, your doctor will discuss other options with you and continue to treat you with the best means available.

You may withdraw your permission to use your personal health information for this study at any time by letting the study doctor know. However, this would also mean that you withdraw from the study. Your study data that was recorded before you withdrew will be used but no information will be collected or sent to the sponsor after you withdraw your permission.

Your rights to privacy are legally protected by federal and provincial laws that require safeguards to ensure that your privacy is respected.

By signing this form you do not give up any of your legal rights against the investigators, sponsor or involved institutions for compensation, nor does this form relieve the investigators, sponsor or involved institutions of their legal and professional responsibilities.

You will be given a copy of this signed and dated consent form prior to participating in this study.

### **CONFLICT OF INTEREST**

Note: Please include details of any actual or potential conflict of interest concerning this study.

This centre is receiving funds from the Canadian Cancer Trials Group to help offset the costs of conducting this research. CCTG is a non-profit research group based on donated support.

The researchers, this centre, and the CCTG will not receive any direct benefit for conducting this study.

# **CONTACTS**

| If you have questions about taking part in this study, or if you suffer a research-related injury, you should talk to your study doctor. Or, you can meet with the doctor who is in charge of the study at this institution. That person is: | |
|---|---|
| Name | Telephone |
| If you have questions about your rights as a participant or about ethical issues related to this study, you can talk to someone who is not involved in the study at all. That person is: | |
| Name | Telephone |

AMEND #1: 2017-FEB-02

# **SIGNATURES**

- All of my questions have been answered,
- I understand the information within this informed consent form,
- I allow access to my medical records and specimens as explained in this consent form,
- I do not give up any of my legal rights by signing this consent form,

| • | I agree to take part in this study | y. | |
|---|---|---|---|
| Si | gnature of Participant | Printed Name | <br>Date |
| | gnature of Person Conducting<br>e Consent Discussion | Printed Name | <br>Date |
| Pa | articipant Assistance | | |
| Co | omplete the following declarati | ion only if the participar | nt is unable to read: |
| • | The informed consent form was accurately explained to, and apparently understood by, the participant, and, | | |
| • | Informed consent was freely given by the participant. | | |
| Si | gnature of Impartial Witness | Printed Name | <br>Date |
| laı | omplete the following declarati<br>nguage in which the consent follows: | | nt has limited proficiency in the pretation was provided as |
| • | The informed consent discussion was interpreted by an interpreter, and, | | |
| • | A sight translation of this document was provided by the interpreter as directed by the research staff conducting the consent. | | |
| In | terpreter declaration and signa | ature: | |
| to | | ovided a sight translation | interpretation for the discussion that of this document as directed by the |
| Si | gnature of Interpreter | Printed Name | <br>Date |